CLINICAL TRIAL: NCT03990610
Title: Assessment of Outcomes Following Prophylactic Lymph Node Transfer in Patients Undergoing Autologous Breast Reconstruction
Brief Title: An Investigational Surgical Procedure (Vascularized Lymph Node Transfer) in Reducing the Risk of Lymphedema in Patients With Breast Cancer Undergoing Breast Reconstruction
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-0528; NCI-2019-03182 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0528 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2019-06-17; First posted 2019-06-19 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-08

CONDITIONS: Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms | interventions — Mammaplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (vascularized lymph node transfer) (Experimental): Patients undergo vascularized lymph node transfer during standard of care breast reconstructive surgery.
  Interventions: Procedure: Mammoplasty; Procedure: Vascularized Lymph Node Transfer

INTERVENTIONS:
Procedure: Mammoplasty — Undergo standard of care breast reconstructive surgery
  Other Names: Breast Reconstruction
Procedure: Vascularized Lymph Node Transfer — Undergo vascularized lymph node transfer
  Other Names: VLNT

SUMMARY:
This trial studies how an investigational surgical procedure called vascularized lymph node transfer works in lowering the risk of arm swelling (lymphedema) in patients with breast cancer undergoing breast reconstruction. Patients who undergo breast reconstruction are often at high risk of developing lymphedema. Vascularized lymph node transfer involves transferring lymph nodes from an unaffected area of the body to replace those removed as part of treatment, which may lower the risk of lymphedema after breast reconstruction.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine incidence of patients who develop lymphedema following autologous breast reconstruction.

SECONDARY OBJECTIVES:

I. Determine the overall complications of prophylactic vascularized lymph node transfers.

II. Compare the incidence of patients who develop lymphedema following autologous breast reconstruction among patients who had prophylactic lymph node transfer and a historical cohort who did not have prophylactic lymph node transfer.

OUTLINE:

Patients undergo vascularized lymph node transfer during standard of care breast reconstructive surgery.

After completion of study, patients are followed up for 3 weeks, at 3 and 6 months, and then at 1 and 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have undergone treatment (mastectomy, axillary lymph node dissection [ALND], radiation and chemotherapy) for breast cancer and are seeking breast reconstruction

Exclusion Criteria:

* Patients that are known to be pregnant at the time of surgery
* Patients with a known hypersensitivity to indocyanine green (ICG) and/or isosulfan blue (Lymphazurin)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-05-24 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Incidence rate of lymphedema development | At 12 months after surgery
  Summary statistics such as means, standard deviations, median and range for continuous variables, and frequencies and percentages for categorical variables will be reported. The rate of lymphedema and its 95% exact confidence interval will be estimated.
Time to lymphedema development | Up to 2 years
  Will be estimated by the Kaplan-Meier method.

SECONDARY OUTCOMES:
Incidence rate of lymphedema development | Up to 2 years
  The incidence of lymphedema between patients who undergo vascularized lymph node transfer (VLNT) and historical cohorts who do not will be compared. The inverse probability of treatment weighting using the propensity scores will be applied to estimate the effect of VLNT.
Complications of prophylactic VLNT | Within 30 days after surgery
  Overall complications will include infections, dehiscence, hematoma, seroma and flap compromises. The 95% exact confidence interval will be estimated.

CONTACTS AND LOCATIONS:
Overall Officials: Edward I Chang, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2022-10-04): https://cdn.clinicaltrials.gov/large-docs/10/NCT03990610/ICF_000.pdf